CLINICAL TRIAL: NCT01953302
Title: Modified "Open Intraperitoneal Mesh" Technique of Incisional Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varazdin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24011983
Record Dates: First submitted 2013-09-21; First posted 2013-09-30 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2017-04

CONDITIONS: Incisional Ventral Hernia; Recurrent Ventral Hernia
Keywords: ventral hernia; infection; hematoma; seroma; recurrence; mesh technique
MeSH Terms: conditions — Hernia, Ventral; Infections; Hematoma; Seroma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- modified "open mesh technique" (Experimental): We performed an "open" intraperitoneal mesh technique in all patients: we placed surgical mesh of appropriate size intraperitoneally with transfascial fixation and drainage.
  Interventions: Procedure: modified "open mesh technique"

INTERVENTIONS:
Procedure: modified "open mesh technique" — We positioned mesh intraperitoneally so it can provide adequate mechanical support to the weakened abdominal wall. We also preserved hernia sack to conceal the mesh.
  Other Names: Proceed Surgical Mesh; VycrilTM,2-0 resorbing sutures

SUMMARY:
Ventral hernias, primary and recurrent, are major surgical challenge. We aim to investigate efficacy of modified technique of ventral hernias repair: an "open intraperitoneal mesh" technique.

DETAILED DESCRIPTION:
We analyzed early postoperative complications (EPCs; wound infection, hematoma, and seroma) and late postoperative complications (recurrence) in 124 patients operated for IHs and recurrent IHs (RIHs) using our new technique. Our technique involved repairing hernias by preserving the hernia sac, which was later used to conceal the mesh that replaced the abdominal wall defect, thus dividing the mesh from subcutaneous tissue.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* American Society of Anesthesiologists physical status I, II, III

Exclusion Criteria:

* refusal of the patients to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranko Stare, MD, PhD, Principal Investigator — Varazdin General Hospital
Locations (1):
- Varazdin General Hospital, Varaždin, Croatia

REFERENCES:
- [Result] Pajtak A, Stare R, Biskup I, Lukic A, Skorjanec S, Hrzenjak K. A modified open intraperitoneal mesh (Garestin) technique for incisional ventral hernia repair. Asian J Surg. 2017 Jul;40(4):278-284. doi: 10.1016/j.asjsur.2016.02.001. Epub 2016 May 18. PMID 27209474

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified "Open Mesh Technique"
Started | 124
Completed | 124
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Modified "Open Mesh Technique"
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 46
Region of Enrollment [Number; unit: participants]
  Croatia | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Early Postoperative Complications (Wound Infections, Seroma, Hematoma)
Description: we counted number of patinetns with wound infection, seroma, hematoma that occured in the early postoperative time
Time Frame: four weeks after the surgery
Measure: Number; unit: participants
Arm/Group | Modified "Open Mesh Technique"
Number analyzed (Participants) | 124
participants
  Infection | 9
  Seroma | 21
  Hematoma | 2
  No complications | 92

2. Secondary Outcome: Number of Patients With Postoperative Hernia Recurrence
Time Frame: up to 36 months after the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Modified "Open Mesh Technique"
Number analyzed (Participants) | 124
Participants
  Reccurence with early complications | 7
  Reccurence with infection | 4
  No reccurence | 113

ADVERSE EVENTS:
Arm/Group | Modified "Open Mesh Technique"
Serious Adverse Events (participants affected / at risk) | 0/124
Other Adverse Events (participants affected / at risk) | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes